CLINICAL TRIAL: NCT03536780
Title: Phase II Trial of Avelumab in Combination With Gemcitabine in Advanced Leiomyosarcoma as a Second-line Treatment
Brief Title: Avelumab in Combination With Gemcitabine in Advanced Leiomyosarcoma as a Second-line Treatment
Acronym: EAGLES
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gachon University Gil Medical Center (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry); Chong Kun Dang Pharmaceutical Corp. (Industry)
Responsible Party: Principal Investigator, Young Saing Kim, Associate Professor, Gachon University Gil Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCSG UN18-06; MS100070_0069 (Other: Merck KGaA)
Record Dates: First submitted 2018-05-10; First posted 2018-05-25 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Leiomyosarcoma Metastatic
MeSH Terms: interventions — avelumab; Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Avelumab and Gemcitabine (Experimental)
  Interventions: Drug: Avelumab and Gemcitabine

INTERVENTIONS:
Drug: Avelumab and Gemcitabine — * Avelumab: 10 mg/kg by IV infusion over 1 hour, every 2 weeks
  * Gemcitabine: 1000 mg/m2 by IV infusion over 30 minutes on Days 1, 8, and 15 of each 28-day cycle

SUMMARY:
A Phase 2 trial of avelumab plus gemcitabine in advanced leiomyosarcoma as a second line treatment

ELIGIBILITY:
Inclusion Criteria:

1. Unresectable, advanced or metastatic histologically confirmed leiomyosarcoma
2. Progression during or after first-line doxorubicin-based chemotherapy (relapse within 6 months of completion of adjuvant/neoadjuvant chemotherapy containing doxorubicin-based regimen could be considered as first-line therapy.)
3. ECOG PS 0-2
4. At least one measurable lesion according to RECIST v1.1
5. Adequate organ function
6. Life expectancy >= 3 months
7. Negative serum or urine pregnancy test at screening for women of childbearing potential

Exclusion Criteria:

1. Prior treatment history of anti-PD-1/PD-L1 or anti-CTLA4 treatment
2. Receipt of 2 or more prior systemic treatments for advanced leiomyosarcoma
3. Active or untreated brain metastases or spinal cord compression
4. Prior treatment with gemcitabine
5. History of major surgery within 4 weeks prior to enrollment
6. Chemotherapy or radiotherapy within 3 weeks prior to the study drug commencement
7. Previous malignant disease other than leiomyosarcoma within the last 5 years with the exception of basal or squamous cell carcinoma of skin or carcinoma in situ (bladder, cervical, colorectal, breast)
8. Pregnant or lactating women
9. HIV, HBV, or HCV infection
10. Severe hypersensitivity or anaphylaxis to monoclonal antibody, or uncontrolled bronchial asthma
11. Current use of immunosuppressive agent (exclusion : less than prednisone 10 mg/day or equivalent)
12. Active autoimmune disease
13. Clinically significant cardiovascular disease
14. Clinically significant interstitial pneumonitis or pulmonary fibrosis
15. Vaccination within 4 weeks of the first dose of avelumab and while on trial is prohibited except for administration of inactivated vaccines

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | 3 years
  response rate according to RECIST v1.1

CONTACTS AND LOCATIONS:
Locations (6):
- South Korea (6):
  - Dong-a University Hospital, Busan
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clark MA, Fisher C, Judson I, Thomas JM. Soft-tissue sarcomas in adults. N Engl J Med. 2005 Aug 18;353(7):701-11. doi: 10.1056/NEJMra041866. No abstract available. PMID 16107623
- [Background] Linch M, Miah AB, Thway K, Judson IR, Benson C. Systemic treatment of soft-tissue sarcoma-gold standard and novel therapies. Nat Rev Clin Oncol. 2014 Apr;11(4):187-202. doi: 10.1038/nrclinonc.2014.26. Epub 2014 Mar 18. PMID 24642677
- [Background] Hensley ML, Maki R, Venkatraman E, Geller G, Lovegren M, Aghajanian C, Sabbatini P, Tong W, Barakat R, Spriggs DR. Gemcitabine and docetaxel in patients with unresectable leiomyosarcoma: results of a phase II trial. J Clin Oncol. 2002 Jun 15;20(12):2824-31. doi: 10.1200/JCO.2002.11.050. PMID 12065559
- [Background] Seddon B, Strauss SJ, Whelan J, Leahy M, Woll PJ, Cowie F, Rothermundt C, Wood Z, Benson C, Ali N, Marples M, Veal GJ, Jamieson D, Kuver K, Tirabosco R, Forsyth S, Nash S, Dehbi HM, Beare S. Gemcitabine and docetaxel versus doxorubicin as first-line treatment in previously untreated advanced unresectable or metastatic soft-tissue sarcomas (GeDDiS): a randomised controlled phase 3 trial. Lancet Oncol. 2017 Oct;18(10):1397-1410. doi: 10.1016/S1470-2045(17)30622-8. Epub 2017 Sep 4. PMID 28882536
- [Background] Pautier P, Floquet A, Penel N, Piperno-Neumann S, Isambert N, Rey A, Bompas E, Cioffi A, Delcambre C, Cupissol D, Collin F, Blay JY, Jimenez M, Duffaud F. Randomized multicenter and stratified phase II study of gemcitabine alone versus gemcitabine and docetaxel in patients with metastatic or relapsed leiomyosarcomas: a Federation Nationale des Centres de Lutte Contre le Cancer (FNCLCC) French Sarcoma Group Study (TAXOGEM study). Oncologist. 2012;17(9):1213-20. doi: 10.1634/theoncologist.2011-0467. Epub 2012 Aug 20. PMID 22907974
- [Background] Dunn GP, Bruce AT, Ikeda H, Old LJ, Schreiber RD. Cancer immunoediting: from immunosurveillance to tumor escape. Nat Immunol. 2002 Nov;3(11):991-8. doi: 10.1038/ni1102-991. PMID 12407406
- [Background] Tawbi HA, Burgess M, Bolejack V, Van Tine BA, Schuetze SM, Hu J, D'Angelo S, Attia S, Riedel RF, Priebat DA, Movva S, Davis LE, Okuno SH, Reed DR, Crowley J, Butterfield LH, Salazar R, Rodriguez-Canales J, Lazar AJ, Wistuba II, Baker LH, Maki RG, Reinke D, Patel S. Pembrolizumab in advanced soft-tissue sarcoma and bone sarcoma (SARC028): a multicentre, two-cohort, single-arm, open-label, phase 2 trial. Lancet Oncol. 2017 Nov;18(11):1493-1501. doi: 10.1016/S1470-2045(17)30624-1. Epub 2017 Oct 4. PMID 28988646
- [Background] Kelly K, Infante JR, Taylor MH, Patel MR, Wong DJ, Iannotti N, Mehnert JM, Loos AH, Koch H, Speit I, Gulley JL. Safety profile of avelumab in patients with advanced solid tumors: A pooled analysis of data from the phase 1 JAVELIN solid tumor and phase 2 JAVELIN Merkel 200 clinical trials. Cancer. 2018 May 1;124(9):2010-2017. doi: 10.1002/cncr.31293. Epub 2018 Feb 22. PMID 29469949
- [Background] Galluzzi L, Senovilla L, Zitvogel L, Kroemer G. The secret ally: immunostimulation by anticancer drugs. Nat Rev Drug Discov. 2012 Feb 3;11(3):215-33. doi: 10.1038/nrd3626. PMID 22301798
- [Background] Chen G, Emens LA. Chemoimmunotherapy: reengineering tumor immunity. Cancer Immunol Immunother. 2013 Feb;62(2):203-16. doi: 10.1007/s00262-012-1388-0. Epub 2013 Feb 7. PMID 23389507
- [Background] Kim JM, Chen DS. Immune escape to PD-L1/PD-1 blockade: seven steps to success (or failure). Ann Oncol. 2016 Aug;27(8):1492-504. doi: 10.1093/annonc/mdw217. Epub 2016 May 20. PMID 27207108